CLINICAL TRIAL: NCT03880968
Title: Treat-to-Target Strategy With Etanercept for Ankylosing Spondylitis: a Prospective, Randomized Multicentric Study on Disease Activity Guided Etanercept Tapering or Discontinuation
Brief Title: Treat-to-Target Strategy With Etanercept for Ankylosing Spondylitis
Acronym: T2TEAS
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Affiliated Hospital of Jiaxing University (Other); Shaoxing Second Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Wenzhou Central Hospital (Other); Zhejiang Provincial People's Hospital (Other); Shaoxing People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-13
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2019-03

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- inactive - half dosage tapering: Active AS patients with AS disease activity score (ASDAS)≥2.1 were recruited from ten hospitals, initially managed with ETN 50mg weekly for 12 weeks, and then randomized into subgroups with different tapering or discontinuation strategies according to ASDAS at week 12. Patients in this arm were those who achieved inactive disease (ASDAS<1.3, group A) at week 12 and assigned to sequential tapering group (A1).
  Interventions: Drug: tapering or discontinuation of etanercept
- inactive - discontinuation: Active AS patients with AS disease activity score (ASDAS)≥2.1 were recruited from ten hospitals, initially managed with ETN 50mg weekly for 12 weeks, and then randomized into subgroups with different tapering or discontinuation strategies according to ASDAS at week 12. Patients in this arm were those who achieved inactive disease (ASDAS<1.3, group A) at week 12 and then assigned to discontinuation group (A2).
  Interventions: Drug: tapering or discontinuation of etanercept
- low disease activity - half dosage tapering: Active AS patients with AS disease activity score (ASDAS)≥2.1 were recruited from ten hospitals, initially managed with ETN 50mg weekly for 12 weeks, and then randomized into subgroups with different tapering or discontinuation strategies according to ASDAS at week 12. Patients in this arm were those who reached low disease activity (LDA) (1.3≤ASDAS<2.1, group B) and designated to sequential tapering group (B1).
  Interventions: Drug: tapering or discontinuation of etanercept
- low disease activity - full dosage tapering: Active AS patients with AS disease activity score (ASDAS)≥2.1 were recruited from ten hospitals, initially managed with ETN 50mg weekly for 12 weeks, and then randomized into subgroups with different tapering or discontinuation strategies according to ASDAS at week 12. Patients in this arm were those who reached low disease activity (LDA) (1.3≤ASDAS<2.1, group B) and designated to delayed tapering group (B2) with extra 12 weeks of full dose ETN.
  Interventions: Drug: tapering or discontinuation of etanercept
- low disease activity - discontinuation: Active AS patients with AS disease activity score (ASDAS)≥2.1 were recruited from ten hospitals, initially managed with ETN 50mg weekly for 12 weeks, and then randomized into subgroups with different tapering or discontinuation strategies according to ASDAS at week 12. Patients in this arm were those who reached low disease activity (LDA) (1.3≤ASDAS<2.1, group B) and designated to discontinuation group (B3).
  Interventions: Drug: tapering or discontinuation of etanercept

INTERVENTIONS:
Drug: tapering or discontinuation of etanercept — Active AS patients initially managed with ETN 50mg weekly for 12 weeks, and then randomized into subgroups with different tapering or discontinuation strategies according to ASDAS at week 12. Patients who achieved inactive disease (ASDAS<1.3, group A) at week 12 were either assigned to sequential tapering group (A1) or discontinuation group (A2), and those who reached low disease activity (LDA) (1.3≤ASDAS<2.1, group B) were designated to sequential tapering group (B1), delayed tapering group (B2) or discontinuation group (B3).
  Other Names: rhTNFR:Fc, Yisaipu

SUMMARY:
Evaluate the disease activity guided tapering and discontinuation strategies of etanercept (ETN) in patients with ankylosing spondylitis (AS) in 48 weeks.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS), a subset of axial spondyloarthritis (axSpA), is a chronic inflammatory disorder characterized by inflammatory back pain and predominant involvement of sacroiliac joints and spine, leading to bony fusion of vertebrae and eventually disability in some patients. Nonsteroidal anti-inflammatory drugs (NSAIDs) are recognized as a first-line therapy for AS, but the overall response rates to NSAIDs are considerably unsatisfactory. With the advent of biologics, the outcomes of AS patients have been greatly improved. Biologics including tumor necrosis factor α (TNFα) inhibitors (TNFi) have been included in many recommendations for the treatment of AS. Etanercept, a recombinant human TNFα receptor, is capable of binding to TNFα and blocking its biological activities. It is effective in relieving symptoms, improving physical function, and reducing disease activity in patients with AS, and generally no severe adverse effects have been reported. However, the high expense of biologics restricts their long-term use, which urges a viable strategy to reduce the dosage of biologics while maintaining an optimal therapeutic efficacy. To investigate the stepwise tapering and discontinuation of TNFi based on disease activity in patients with AS, a 48-week, prospective, randomized, multicentric study was conducted. An etanercept biosimilar, rhTNFR:Fc (recombinant TNF receptor: Fc fusion protein, Yisaipu), which is one of the most widely used biosimilars in China, was used in this study.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 years old and 65 years old with AS, according to 1984-revised New York classification criteria.
* an active disease of ASDAS with C reactive protein (ASDAS-CRP) ≥2.1.
* a disease duration of 6 months to 30 years.
* no exposure to biologics in recent 6 months before recruitment. Concomitant medications with NSAIDs, conventional disease modifying anti-rheumatic drugs (cDMARDs), or prednisone or a prednisone equivalent (≤10mg/day), were allowed to continue if they were maintained at a stable dose for 4 weeks or more from baseline.

Exclusion Criteria:

* late-stage patients with spinal fusion.
* patients with severe cardiac, hepatic, renal, hematologic or endocrine diseases.
* patients with a history of multiple sclerosis, current or past malignancy.
* patients who were pregnant, or planning to become pregnant, or breastfeeding.
* patients with active or recurrent infections, or those who required oral antibiotics 2 weeks or intravenous antibiotics 4 weeks before screening.
* patients with current or past or potential tuberculosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AS were recruited in this study. Eligible patients were aged between 18 years old and 65 years old, and were diagnosed with AS according to 1984 revised New York classification criteria. Only patients meet both inclusion and exclusion criteria were included.
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Cumulative flare rates at week 48 with different tapering or discontinuation strategies | 48 weeks
  Cumulative flare rates at week 48 with different tapering or discontinuation strategies

CONTACTS AND LOCATIONS:
Overall Officials: Huaxiang Wu, Principal Investigator — wuhx8855@sina.com

REFERENCES:
- [Derived] Zhang T, Zhu J, He D, Chen X, Wang H, Zhang Y, Xue Q, Liu W, Xiang G, Li Y, Yu Z, Wu H. Disease activity guided stepwise tapering or discontinuation of rhTNFR:Fc, an etanercept biosimilar, in patients with ankylosing spondylitis: a prospective, randomized, open-label, multicentric study. Ther Adv Musculoskelet Dis. 2020 Jun 2;12:1759720X20929441. doi: 10.1177/1759720X20929441. eCollection 2020. PMID 32536984